CLINICAL TRIAL: NCT03151252
Title: Improvement of Foodallergy Diagnostic in Gastrointestinal Tract With a New Kind of Sampling
Brief Title: Improvement of Foodallergy Diagnostic in Gastrointestinal Tract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Foodallergy in Colon
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Food allergy (Other): Patients with confirmed foodspecific- IgE antibodies in blood
  Interventions: Diagnostic Test: Cytobrush
- healthy controls (Other): participants without foodspecific- IgE antibodies in blood and other gastrointestinal symptoms
  Interventions: Diagnostic Test: Cytobrush
- gastointestinal symptoms without foodallergy in blood (Other): Patients without foodspecific- IgE antibodies in blood, but with gastrointestinal symptoms
  Interventions: Diagnostic Test: Cytobrush

INTERVENTIONS:
Diagnostic Test: Cytobrush — During the endoscopic Investigation the mucosa cells were collected by brushing the colon via cytobrush.

SUMMARY:
Currently, diagnostic possibilities for the detection of food allergy in the gastrointestinal tract are scarce. The endoscopic segmental Lavage is the method of choice, but it´s controversial.

Additional to the endoscopic segmental lavage fluid a cytobrush is used for collecting the mucosa cells and biopsies are taken. Comparative to the Lavage specific IgE antibodies, Tumor necrosis factor- alpha, Eosinophilic cation protein and mastcell tryptase were measured.

ELIGIBILITY:
Inclusion Criteria:

* all patients with suspicion of food intolerance and confirmed food allergy

Exclusion Criteria:

* pregnant and patients under allergy medication (antihistaminic, cortison)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
detection of specific IgE Antibodies in colon | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports, Friedrich-Alexander-University Erlangen-Nuremberg, Erlangen, Germany

REFERENCES:
- [Derived] Dieterich W, Tietz E, Kohl M, Konturek PC, Rath T, Neurath MF, Zopf Y. Food Intolerance of Unknown Origin: Caused by Mucosal Inflammation? A Pilot Study. Clin Transl Gastroenterol. 2021 Feb 17;12(2):e00312. doi: 10.14309/ctg.0000000000000312. PMID 33600102